CLINICAL TRIAL: NCT05807243
Title: Descriptive Study of Molecular Markers of Immunosenescence With Nutritional Intervention to Evaluate the Implementation of Digital Tools in the Capture of Nutritional Data
Brief Title: Description of Immunosenescence Biomarkers and Nutritional Intervention to Evaluate the Implementation of Digital Tools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMDEA Food (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IMD: PI-052
Record Dates: First submitted 2023-02-27; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Chronic Disease
Keywords: Artificial Intelligence; Multi-modal learning; Nutrition; Biomarkers; Precision Nutrition; Immunosenescence
MeSH Terms: conditions — Chronic Disease | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Traditional → Digital) (Experimental): Participants in both groups will be monitored for a month while following an hypocaloric diet for healthy weight-loss.
  The first group (n=50) will start collecting data via questionnaires (traditional method) for the first two weeks, and switch to the digital data-collection method for the last two weeks.
  Interventions: Other: Dietary intervention for healthy weight loss
- Group 2 (Digital → Traditional) (Experimental): Participants in both groups will be monitored for a month while following an hypocaloric diet for healthy weight-loss.
  The second group (n=50) will start with the digital data-collection method for the first two weeks and switch to the data collection via questionnaires (traditional method) for the last two weeks.
  n=100)
  Interventions: Other: Dietary intervention for healthy weight loss
- Group 3 - Young healthy population (No Intervention): n=100) Descriptive part: Data capture (clinical, anthropometric, lifestyle, genetic, biochemical, metabolomic and lipidomic data, among others) and comparison with the other groups.
- Group 4 - Senior population (No Intervention): n=100) Descriptive part: Data capture (clinical, anthropometric, lifestyle, genetic, biochemical, metabolomic and lipidomic data, among others) and comparison with the other groups.
- Group 5 - Oncological population (No Intervention): (n=100) Descriptive part: Data capture (clinical, anthropometric, lifestyle, genetic, biochemical, metabolomic and lipidomic data, among others) and comparison with the other groups.
- Group 6 - COVID-19 population (No Intervention): (n=100) patients who developed severe forms of COVID-19 or persistent COVID-19. Descriptive part: Data capture (clinical, anthropometric, lifestyle, genetic, biochemical, metabolomic and lipidomic data, among others) and comparison with the other groups.

INTERVENTIONS:
Other: Dietary intervention for healthy weight loss — Balanced and varied dietary plan adjusted to each participant's needs, with an approximate reduction of 500 Kcal from their total metabolic expenditure. The diet will be followed by the subjects during the 4 weeks of the study.
  Arms: Group 1 (Traditional → Digital); Group 2 (Digital → Traditional)

SUMMARY:
Descriptive comparative study of immunosenescence markers and their association with nutritional, metabolic, metabolomic and genetic characteristics in young (control), senior (age-associated immunosenescence), and populations susceptible to premature immunosenescence such as obese patients, cancer patients and patients who developed severe forms of COVID19 or persistent COVID19.

In one of these populations of premature immunosenescence, the population group with overweight or obesity, a prospective and cross-sectional nutritional intervention study is proposed, with data capture and monitoring using digital tools, to evaluate the evolution of immunosenescence markers and assess more objectively and effectively the nutritional status and help in making personalised decisions thanks to the application of these tools. This nutritional intervention will be focused on controlled and safe weight loss that will allow the capture of a large number of variables on lifestyle and dietary habits, nutritional assessment, biochemical, metabolic, genetic, metagenomic, lipidomic and metabolomic markers measured statically and also continuously.

DETAILED DESCRIPTION:
The study consists of data capturing to evaluate the differential pattern of molecular markers of immunosenescence in different population groups, and applying a hypocaloric diet in the obesity subgroup together with recommendations for improving lifestyle habits. The data capture of this group during the intervention will be carried out with different sensors and questionnaires for a month. To do this, they will have to follow the explanations of the researchers.

The data capture during the nutritional intervention (only for the overweight and obese population group) will be done as follows:

Group 1 (Traditional → Digital): will start with traditional data-collection methods, i.e. filling in nutritional and lifestyle questionnaires (Visit 1 to Visit 2). After two weeks, they will start capturing data digitally through the application of sensors (Visit 2 to Visit 3).

Group 2 (Digital → Traditional): will start with digital data-collection methods, using sensors and taking pictures of what they eat with a smartphone (Visit 1 to Visit 2). After two weeks, they will start capturing data traditionally, by filling in nutritional and lifestyle questionnaires (Visit 2 to Visit 3).

The nutritional intervention participant group will follow the tailored nutritional weight loss diet and lifestyle guidelines, which will be provided to them at the start of the study by the researchers. In addition, they should follow instructions for proper continuous data collection using sensors. This will avoid biases in the data collection process.

ELIGIBILITY:
Inclusion Criteria (commun for all groups):

* Men/women
* Minimum 18 years old
* Adequate cultural level and understanding of the clinical study.
* Agree to participate voluntarily in the study and give written informed consent.

Population-specific inclusion criteria:

* Overweight/obese population:

  * BMI 25-35 Kg/m2
  * Ability to handle electronic devices for data capture.
* Healthy young population:

  * Between 18 and 25 years old (both inclusive).
* Senior population

  * Over 55 years of age.
* Oncology patients

  * Over 18 years of age.
  * With a clinical diagnosis of an active tumour process.
* Patients who developed severe or persistent COVID-19:

  * Severe COVID-19: Patients who have suffered from COVID-19 disease and whose symptomatology is considered within the clinical pictures of severity of this disease, which may include: severe pneumonia, acute respiratory distress syndrome (ARDS), presence of respiratory failure (SaO2 <90% room air) or respiratory rate ≥ 30 breaths per minute, sepsis, septic shock, thromboembolism and multi-organ dysfunction (including acute cardiac and renal injuries).
  * COVID-19 persistence: Patients who have had COVID-19 disease and who remain with active symptomatology after what is considered the acute phase of the disease, after 4 or even 12 weeks, with symptoms persisting over time.

Exclusion Criteria:

* Dementia, mental illness or diminished cognitive function that can hinder the subject's participation on the study.
* Severe diseases (liver disease, kidney disease, etc.)
* BMI > 35 Kg/m2
* Pregnancy or breastfeeding.

Population-specific exclusion criteria:

* Overweight/obese population:

  * BMI <25 Kg/m2 or > 35 Kg/m2
  * Pharmacological treatment for weight loss.
  * Refusal to be monitored for one month by means of sensors and nutritional visits.
  * Refusal to follow healthy eating guidelines for weight loss.
* Healthy young population:

  * Chronic or acute pathologies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
BMI | 1 month
  Only in the obese/overweight population.
  Change in body mass index (Kg/m2)
Blood Glucose | 1 month
  Change in blood glucose (mg/dl). Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Concentration of interstitial glucose | 15 days
  Only in the obese/overweight population.
  Change in Interstitial Glucose (mgl/dl) measured continuously with the Freestyle glucometer (Abbott Laboratories)
Blood lymphocytes | 12 months
  Variation in the percentage of blood lymphocytes analysed by flow cytometry in five different population groups (young healthy population, elderly, overweight-obese, cancer patients, and patients who developed severe forms of COVID-19 or persistent COVID-19).
  Other variables (described in the Secondary Outcomes), such as biochemical parameters, genetical data, microbiota, etc., will also be analyzed in order to identify specific molecular markers of immunosenescence.

SECONDARY OUTCOMES:
Weight | 1 month
  Weight change (Kg)
WC | 1 month
  Change in waist circumference (cm)
Body composition | 1 month
  Change in % of fat mass
Blood pressure | 1 month
  During the 2 weeks in which the participant gathers the information via Traditional data-collection method, it will be measured in the study visits with an automatic Digital Blood Pressure Monitor Model M3 (OMRON HEALTHCARE UK, Kyoto, Japan).
  And during the 2 weeks in which the participant gathers the information via the Digital data-collection method, it will be measured with the Smartwatch Fitbit Sense.
Heart Rate | 1 month
  During the 2 weeks in which the participant gathers the information via Traditional data-collection method, it will be measured in the study visits with an automatic Digital Blood Pressure Monitor Model M3 (OMRON HEALTHCARE UK, Kyoto, Japan).
  And during the 2 weeks in which the participant gathers the information via the Digital data-collection method, it will be measured with the Smartwatch Fitbit Sense.
Dietary intake | 1 month
  Traditional data-collection method: Two 3-day dietary records (for two working days and a holiday); Digital data-collection method: Pictures of food taken with a smartphone.
Physical activity | 1 month
  One same outcome measured during 2 weeks with one method and during the other 2 weeks with another method:
  During the 2 weeks in which the participant gathers the information via Traditional data-collection method, it will be measured via the validated International Physical Activity Questionnaire (USA Spanish version translated 3/2003 - Short last 7 DAYS self-administered version of the IPAQ - Revised August 2002).
  And during the 2 weeks in which the participant gathers the information via the Digital data-collection method, it will be measured with the Smartwatch Fitbit Sense.
Sleep | 1 month
  One same outcome measured during 2 weeks with one method and during the other 2 weeks with another method:
  During the 2 weeks in which the participant gathers the information via Traditional data-collection method, it will be measured via the validated Oviedo Sleep Questionnaire. In the Oviedo Sleep Questionnaire, the higher the score, the greater insomnia's severity.
  And during the 2 weeks in which the participant gathers the information via the Digital data-collection method, it will be measured with the Smartwatch Fitbit Sense.
Mental health state | 1 month
  One same outcome measured during 2 weeks with one method and during the other 2 weeks with another method:
  During the 2 weeks in which the participant gathers the information via Traditional data-collection method, it will be measured via the validated Depression Anxiety and Stress Scale - 21 (DASS-21). In the Depression Anxiety and Stress Scale, the higher the score, the greater the stress, anxiety and depression levels.
  And during the 2 weeks in which the participant gathers the information via the Digital data-collection method, it will be measured with the Smartwatch Fitbit Sense.
Cognition | 1 month
  Measured via the validated Mini-mental state examination (MMSE). In the Mini-mental state examination, the higher the score, the better the cognitive status.
Health status and quality of life | 1 month
  Measured via the validated Short Form-36 Health Survey (SF-36). In the Short Form-36 Health Survey, the higher the score, the better the quality of life and health status.
Percentage of glycated haemoglobin | 1 month
  During the 2 weeks in which the participant gathers the information via Traditional data-collection method, it will be only measured in the study visits with the blood tests.
  And during the 2 weeks in which the participant gathers the information via the Digital data-collection method, it will be measured continuously with the Freestyle glucometer (Abbott Laboratories), and in the study visits with the blood tests.
Total cholesterol | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Low density lipoprotein (LDL) | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
High density lipoprotein (HDL) | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Triglycerides | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Apo A1 | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Apo B | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Insulin | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Glycated hemoglobin (HbA1c) | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Homeostatic model assessment (HOMA) | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Albumin | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Prealbumin | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
C-reactive protein (CRP) | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Leptin | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Adinopectin | 1 month
  Blood samples are going to be collected in visit 1 and visit 3 in the obese population, and in the visit 1 in the other populations.
Faecal microbiota | 1 month
  Faecal microbiota taxonomic profiling through shotgun sequencing.
Gut dysbiosis | 1 month
  Lipopolysaccharide-binding protein (LBP) levels as an indirect measure of intestinal dysbiosis.
Genotype | 1 month
  Genotyping of single nucleotide genetic variants (SNPs) and specific mutations associated with metabolism, nutrition and immunodegenerative processes.
Gene expression | 1 month
  Expression panels in genes related to the regulation of metabolism, inflammation, immunity, oxidation, nutrition and immunodegenerative processes.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Ramírez de Molina, PhD, Principal Investigator — Fundación IMDEA Alimentación; Enrique Carrillo de Santa Pau, PhD, Principal Investigator — Fundación IMDEA Alimentación; María Isabel Espinosa Salinas, PhD, Principal Investigator — Fundación IMDEA Alimentación; Cristina María Fernández Díaz, PhD, Principal Investigator — Fundación IMDEA Alimentación
Locations (1):
- IMDEA Food, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fontana L, Partridge L. Promoting health and longevity through diet: from model organisms to humans. Cell. 2015 Mar 26;161(1):106-118. doi: 10.1016/j.cell.2015.02.020. PMID 25815989
- [Background] GBD 2017 Diet Collaborators. Health effects of dietary risks in 195 countries, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 May 11;393(10184):1958-1972. doi: 10.1016/S0140-6736(19)30041-8. Epub 2019 Apr 4. PMID 30954305
- [Background] Moore JB. From personalised nutrition to precision medicine: the rise of consumer genomics and digital health. Proc Nutr Soc. 2020 Aug;79(3):300-310. doi: 10.1017/S0029665120006977. Epub 2020 May 29. PMID 32468984
- [Derived] Lacruz-Pleguezuelos B, Bazan GX, Romero-Tapiador S, Freixer G, Tolosana R, Daza R, Fernandez-Diaz CM, Molina S, Crespo MC, Laguna T, Marcos-Zambrano LJ, Aguilar-Aguilar E, Fernandez-Cabezas J, Cruz-Gil S, Fernandez LP, Vera-Rodriguez R, Fierrez J, Ramirez de Molina A, Ortega-Garcia J, Morales A, Carrillo de Santa Pau E, Espinosa-Salinas I. AI4Food, a feasibility study for the implementation of automated devices in the nutritional advice and follow up within a weight loss intervention. Clin Nutr. 2025 May;48:80-89. doi: 10.1016/j.clnu.2025.03.003. Epub 2025 Mar 11. PMID 40168934
- See also: Research team profile — https://www.food.imdea.org/research/precision-nutrition-programs/program-cancer
- See also: Research team profile — https://www.food.imdea.org/computational-biology
- See also: Research team profile — https://www.food.imdea.org/services/Platform-Clinical-Trials-Nutrition-and-Health